CLINICAL TRIAL: NCT05612984
Title: Calcium Aspirin Multiple Micronutrients (CAMMS) or Iron-folic Acid (IFA) to Reduce Preterm Birth
Brief Title: Calcium Aspirin Multiple Micronutrients (CAMMS) to Reduce Preterm Birth
Acronym: CAMMS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study grant canceled by donor
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Aga Khan University (Other); Institut Africain de Sante Publique (Unknown); Zvitambo Institute for Maternal and Child Health Research (Unknown); Christiana Care Health Services (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INV-036663
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Preterm Labor; Small for Gestational Age at Delivery; Hypertensive Disorder of Pregnancy; Low Birth Weight; Neonatal Death
MeSH Terms: conditions — Obstetric Labor, Premature; Toxemia; Perinatal Death

STUDY DESIGN:
Intervention Model Description: Pregnant women will be individually randomized to daily CAMMS or IFA from recruitment (at 6<20 weeks gestation) to delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium aspirin multiple micronutrients (Experimental): 500 mg elemental calcium (as 1250 mg calcium carbonate) 81 mg aspirin
  1 tablet United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) formula, which is a Multiple Micronutrient Supplement (MMS) for pregnant women
  Interventions: Combination Product: Calcium aspirin multiple micronutrients
- Iron folic acid (Active Comparator): 60 mg iron + 400 μg folic acid given as a combined tablet
  Interventions: Dietary Supplement: Iron-folic Acid

INTERVENTIONS:
Combination Product: Calcium aspirin multiple micronutrients — Women randomized to CAMMS will receive weekly blister cards containing all 3 components: 1 81 mg aspirin tablet, 1 UNIMMAP MMS, and 1 500-mg elemental calcium tablets. Blister packages will be labeled with times of day and days of week when tablets are to be taken. 4 weekly blister cards will be packaged in one unit box.
  Other Names: CAMMS
  Arms: Calcium aspirin multiple micronutrients
Dietary Supplement: Iron-folic Acid — Women randomized to IFA will receive monthly (28-day) blister cards containing containing 1 combined IFA tablet to be taken each day. 1 4-weekly blister card will be packaged in one unit box.
  Other Names: IFA
  Arms: Iron folic acid

SUMMARY:
This trial will evaluate the impact of an integrated intervention of daily maternal calcium, aspirin, and multiple micronutrients (CAMMS) compared to iron-folic acid (IFA) during pregnancy on preterm birth and other adverse birth outcomes. Both interventions will be delivered through existing antenatal service platforms using context-specific strategies informed by formative research incorporating human-centered design processes to achieve high acceptability and high adherence, in three low-income countries with diverse contexts: Burkina Faso, Pakistan, and Zimbabwe.

DETAILED DESCRIPTION:
The CAMMS trial is an individually randomized, unblinded, phase III trial comparing aspirin, calcium and multiple micronutrients (intervention) versus iron-folic acid (control) among 10,000 pregnant women. The primary outcome is total preterm birth, stratified by spontaneous and indicated. Eligible pregnant women will be enrolled from antenatal clinics in three study populations in Burkina Faso, Pakistan, and Zimbabwe following written informed consent.

All women attending antenatal care (ANC) who are positive on a urine pregnancy test and have a fetal ultrasound examination confirming fetal heartbeat, intrauterine pregnancy, and gestational age 6<20 weeks' will be eligible for enrollment. Women who are <6 weeks will be rescheduled for 2-3 weeks later. Baseline data and clinical assessments will be conducted, and women will be randomized to daily ingestion of CAMMS or IFA until delivery. In Burkina Faso, for women randomized to CAMMS, the aspirin will be withheld until 13 weeks' gestation when it can be initiated concurrently with sulfadoxine-pyrimethamine. Women will receive context-specific adherence promotion interventions designed during formative research incorporating Human-Centered Design (HCD) processes in each country. Mothers will be followed up at 4-weekly intervals throughout pregnancy plus an additional study contact (by visit, phone call, WhatsApp, or text message) at 1-2 weeks after starting the study drug to check for tolerance and adherence. Women may also be seen at closer intervals in the third trimester by the Ministry of Health clinics. Women will be encouraged to deliver in a health institution.

Between baseline and delivery, research procedures will be undertaken by research staff based at antenatal clinics during mothers' routine antenatal visits to reduce time burden on participants. Depending on gestational age at recruitment, women will receive 7-11 research visits. One additional visit or contact by text-message (SMS) or phone call will occur one-two weeks after randomization to check that the women is tolerating and correctly taking the interventions.

At delivery, infant weight and gestational age will be measured/determined by research staff based at delivery clinics or, for home deliveries, during home visits conducted within 72 hours of delivery. For infants born outside the study area or who are not reached by research staff within 72 hours, date of birth and birth weight will be transcribed from the infant's health record with source of information noted. In unusual situations where the mother and infant cannot be reached in person before 180 days postpartum but can be reached by telephone, WhatsApp, or Text message, maternal report of data of birth and birth weight will be recorded with the source of information noted. For all infants reached by a research staff member within 72 hours of birth, birth length and head circumference will be measured by standardized research staff with high quality equipment (length measured to nearest 0.1cm with infant length board and Shorr insert-tape (Weigh & Measure LLC., Olney, MD, USA). Mothers and infants will be followed to 42 days post-partum for vital status and post-partum maternal Adverse Events (AEs) and Serious Adverse Events (SAEs). This visit may be conducted in person, by telephone, WhatsApp or text message with the source of information recorded.

ELIGIBILITY:
Inclusion Criteria:

* Woman, confirmed pregnant by urinary pregnancy test
* 6<20 weeks' gestation determined by fetal ultrasound exam;
* Pregnancy must be intrauterine; multiple fetus pregnancies are eligible.
* Women must be willing and able to give informed consent;
* willing to receive antenatal visits at one of the study clinics.
* In Burkina Faso, women must be willing to take monthly sulfadoxine-pyrimethamine.

Exclusion Criteria:

* Pregnant women who are currently taking aspirin, calcium, or MMS;
* have a history of peptic ulcer or have any other contraindications to any of the study drugs;
* have acute or chronic condition that might interfere with the study as judged by the research clinician including severe anemia defined as Hb<5 g/dL;
* have other reasons which, at the study research physician's discretion, mean that receipt of the study drugs or participation in the trial would not be advisable.

NOTE: Women who have been started on IFA by MoH or private health care provider but are willing discontinue the IFA dispensed by MoH and to be randomized to IFA or CAMMS will not be excluded.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total preterm birth | At birth
  Gestational age at birth < 37 weeks, stratified by spontaneous and indicated.

SECONDARY OUTCOMES:
Total very early preterm birth | At birth
  gestational age at birth ≥20 and <28 weeks, stratified by spontaneous and indicated.
Total early preterm birth | At birth
  gestational age ≥28 and <34 weeks, stratified by spontaneous and indicated.
Low birth weight | At birth
  <2500 g
Very low birth weigh | At birth
  <1500 g
Small for gestational age | At birth
  <10th percentile weight for gestational age using INTERGROWTH 21st Reference standards
Stillbirth | Day of fetal loss from > 20 weeks gestation to birth
  fetal loss > 20 gestational weeks
Neonatal death | Day of death, between birth and <28 completed days of life
  death of a live-born infant <28 completed days of life
Miscarriage | Day of fetal loss, up to < 20 weeks gestation
  fetal loss <20 gestational weeks
Live-or-stillbirth-preterm-deliveries | Day of fetal loss or birth, up to < 37 weeks gestation
  stillbirths delivered <37 weeks' gestation + preterm births
Hypertensive disorder of pregnancy | From enrollment at 6<20 weeks gestation through 42 days postpartum
  Maternal Systolic BP>140 and/or Diastolic BP>90 between enrollment and 42 days postpartum
Maternal anemia | 30 weeks' gestation
  Hb<110 g/L during the third trimester of pregnancy
Maternal death | day of woman's death between enrollment at 6<20 weeks gestation up to 42 days postpartum
  death of a woman between enrollment at 6<20 weeks gestation and 42 days postpartum
Perinatal mortality | fetal loss or infant death <28 days of completed life
  Stillbirths + neonatal deaths
Birth weight | At birth
  infant weight (g) ≤ 72 h of birth
Gestational age at birth | At birth
  Completed days of gestation at birth
Weight-for-gestational-age-Z-score at birth | At birth
  WAZ, using INTERGROWTH 21st Reference standards

OTHER OUTCOMES:
Infant birth length and birth head circumference | birth
  Among infants assessed <72 hours after birth by research staff
Tolerance of CAMMS compared to IFA | Up to 42 days post-partum
  Rates of Grade 1 or 2 nausea, vomiting, rash/hives, diarrhea, constipation, and vaginal bleeding from initiation of the interventions through 42 days post-partum
Safety of CAMMS compared to IFA | Up to 42 days post-partum
  Rates of SAEs, Grade 3 or 4 nausea, vomiting, rash/hives, diarrhea, constipation, and vaginal bleeding, stratified by relatedness to the intervention from initiation of the interventions through 42 days post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Jean Humphrey, ScD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Yes
We will deposit anonymized data in an existing repository after publication of the primary and key secondary findings. (
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: About 2 years after the end of the trial when primary and secondary outcomes have been reported in the peer reviewed literature.